CLINICAL TRIAL: NCT02273856
Title: Prospective Multicentre Observational Registry Of Treatments And Outcomes In Patients With Chronic Lymphocytic Leukaemia Or Indolent Non Hodgkin's Lymphoma
Brief Title: Multicentre Registry of Treatments and Outcomes in Patients With Chronic Lymphocytic Leukaemia (CLL) Or Indolent Non Hodgkin's Lymphoma (iNHL)
Acronym: NADIR
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to insufficient subject enrollment and very slow enrollment.
Sponsor: Astellas Pharma International B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: ONC-MA-1002
Record Dates: First submitted 2014-09-02; First posted 2014-10-24 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Indolent Non Hodgkin's Lymphoma (iNHL); Chronic Lymphocytic Leukaemia (CLL)
Keywords: Chronic Lymphocytic Leukaemia (CLL); Indolent Non Hodgkin's Lymphoma (iNHL)
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Treatment naïve patients with CLL
- Treatment naïve patients with iNHL
- Relapsed/refractory patients with CLL
- Relapsed/refractory patients with iNHL

SUMMARY:
The purpose of this study is to document the pharmacological treatment strategies used in treatment naïve and previously treated relapsed/refractory iNHL/CLL patients in the Middle East and North African (MENA) region. This study will also record encountered tumor subtype and stage and the instituted pharmacological treatments, as well as assess the clinical outcomes of treatments.

DETAILED DESCRIPTION:
Patients will be followed up to 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* CLL patients or
* iNHL patients
* Clinical decision made to initiate or adapt treatment of CLL/iNHL("Need to treat")

Exclusion Criteria:

* Patient deemed unfit for enrollment by the documented opinion of the investigator
* Watch and wait patients
* Richter's transformation
* Patients otherwise not eligible for (pharmacological) intervention
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are from the MENA region, and will be selected from sites that are considered clinical centres of excellence in the region.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on different types of pharmacological regimen for treatment of Chronic Lymphocytic Leukaemia (CLL) or Indolent Non Hodgkin's Lymphoma (iNHL) | Baseline, 1 year and 2 years after baseline (up to 30 months)
  Types of combination treatment (including but not limited to R-CHOP [rituximab, cyclophosphamide, vincristine, doxorubicin, prednisone] , FCR [fludarabine, cyclophosphamide, rituximab], COP [cyclophosphamide, doxorubicin, prednisone], BR [bendamustine, rituximab], etc.) will be collected in treatment-naïve and relapsed patients. Data to be described as percentage of patients on each regimen.

SECONDARY OUTCOMES:
Duration of response | up to 30 months
Overall survival | up to 30 months
Progression free survival | up to 30 months
Number of subjects in complete remission | up to 30 months
Number of subjects in partial remission | up to 30 months
Disease type and staging | up to 30 months
Clinical responses | up to 30 months
  Relapses, response or non-response to treatment
Safety as assessed by adverse events | up to 30 months
CLL specific variable: Histology | up to 30 months
  Proportion of different subtypes in CLL: (1) histologically indolent CLL (HIC), defined as morphologically typical CLL with no histologic features of progression or transformation such as increased large cells, large confluent proliferation centers, or high proliferation rate; (2) CLL with histological features of intermediate aggressiveness histologically aggressive CLL [HAC]) (3) Richter's syndrome. Data to be described as percentage.
iNHL specific variables: Histology | up to 30 months
  Proportion of different subtypes in iNHL will be presented. Data to be described as percentage.
Health-related quality of life variables | up to 30 months
  Using EQ-5D questionnaire, including a visual analog scale (dimensions): mobility, self-care, usual activities, pain/discomfort, anxiety/depression
CLL specific variable: Rai/Binet staging systems | up to 30 months
  Percentage of patients in the different stages.
CLL specific variable: Clinically relevant biomarker status | up to 30 months
  Includes immunoglobulin heavy chain variable (IgHV) status, ZAP-70 (70-kDa zeta-associated protein), receptor status (including CD20), cytogenetics (6q, 11q, 13q, and 17p deletion or monosomy, trisomy 12 ). Percentages will be presented for the clinically relevant biomarker status.
iNHL specific variables: Ann Arbor staging classification | up to 30 months
  Percentage of patients in the different stages.
iNHL specific variables: Clinically relevant biomarker status | up to 30 months
  Includes receptor status (including CD20). Percentages will be presented for the clinically relevant biomarker status.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma International B.V.
Locations (8):
- Site JO96201 King Abdullah University Hospital, Irbid, Irbid Governorate, Jordan
- Site KW96501 Kuwait Cancer Control Center, Ash Shuwaykh, Shuwaikh, Kuwait
- Lebanon (2):
  - Site Hammoud Hospital University Medical Center, Beirut, Beyrouth
  - Site Hotel Dieu De France, Beirut, Beyrouth
- Site OM96801 Sultan Qaboos University Hospital, Muscat, Muḩāfaz̧at Masqaţ, Oman
- Site Hamad Medical Coorporation, National Center for Cancer Care and Research, Al Amal Hospital, Doha, Baladīyat ad Dawḩah, Qatar
- Site SA96601 Aseer Central Hospital, Abhā, 'Asir Region, Saudi Arabia
- Site AE97101 Sheikh Khalifa Medical City, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates